CLINICAL TRIAL: NCT06158841
Title: A Phase 3, Multicenter, Randomized, Open Label Study of Etentamig Compared With Standard Available Therapies in Subjects With Relapsed or Refractory Multiple Myeloma (3L+ RRMM Monotherapy Study)
Brief Title: Study Assessing Activity of Intravenous (IV) Etentamig Monotherapy Versus Standard Available Therapies in Adult Participants With Relapsed or Refractory Multiple Myeloma
Acronym: CERVINO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M22-574; 2023-506668-15-00 (Other: EU CT)
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Cervino; Multiple Myeloma; Etentamig; Carfilzomib; Pomalidomide; Elotuzumab; Selinexor; Bortezomib; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; pomalidomide; elotuzumab; selinexor; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Available Therapy (SAT) (Experimental): Participants will receive SAT, in accordance with the local (or applicable) approved label, package insert, summary of product characteristics, and/or the institutional guidelines, as applicable. SAT choices are carfilzomib + dexamethasone (Kd), elotuzumab + pomalidomide + dexamethasone (EloPd), selinexor + bortezomib + dexamethasone (SVd).
  Interventions: Drug: Carfilzomib; Drug: Pomalidomide; Drug: Elotuzumab; Drug: Selinexor; Drug: Bortezomib; Drug: Dexamethasone
- Etentamig (Experimental): Participants will receive etentamig as a monotherapy.
  Interventions: Drug: Etentamig

INTERVENTIONS:
Drug: Etentamig — Intravenous (IV) Infusion
  Other Names: ABBV-383
  Arms: Etentamig
Drug: Carfilzomib — IV Infusion
  Arms: Standard Available Therapy (SAT)
Drug: Pomalidomide — Oral Capsule
  Arms: Standard Available Therapy (SAT)
Drug: Elotuzumab — IV Infusion
  Arms: Standard Available Therapy (SAT)
Drug: Selinexor — Oral Tablet
  Arms: Standard Available Therapy (SAT)
Drug: Bortezomib — Subcutaneous or IV Injection
  Arms: Standard Available Therapy (SAT)
Drug: Dexamethasone — Oral Tablet or IV Infusion
  Arms: Standard Available Therapy (SAT)

SUMMARY:
Multiple myeloma (MM) is a cancer of the blood's plasma cells. The cancer is typically found in the bones and bone marrow (the spongy tissue inside of the bones) and can cause bone pain, fractures, infections, weaker bones, and kidney failure. Treatments are available, but MM can come back (relapsed) or may not get better (refractory) with treatment. This is a study to determine change in disease symptoms of etentamig compared to standard available therapies in adult participants with relapsed/refractory (R/R) MM.

Etentamig is an investigational drug being developed for the treatment of R/R MM. This study is broken into 2 Arms; Arm A and Arm B. In Arm A, participants will receive etentamig as a monotherapy. In Arm B, participants will receive the standard available therapy (SAT) identified by the Investigator during screening, in accordance with the local (or applicable) approved label, package insert, summary of product characteristics, and/or the institutional guidelines, as applicable. Around 380 adult participants with relapsed/refractory multiple myeloma will be enrolled at approximately 140 sites across the world.

In Arm A participants will receive etentamig as an infusion into the vein in 28 day cycles, during the 3.5 year study duration. In Arm B, participants will receive the SAT identified by the Investigator during screening, in accordance with the local (or applicable) approved label, package insert, summary of product characteristics, and/or the institutional guidelines, as applicable, during the 3.5 year study duration.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance of <= 2.
* Diagnosis of relapsed/refractory (R/R) multiple myeloma (MM) during or after the participant's last treatment as stated in the protocol.
* Must have measurable disease with at least 1 of the following assessed within 28 days of enrollment:

  * Serum M-protein >= 0.5 g/dL (>= 5 g/L).
  * Urine M-protein >= 200 mg/24 hours.
  * In participants without measurable serum or urine M protein, serum free light chain (FLC) >= 100 mg/L (10 mg/dL) (involved light chain)and an abnormal serum kappa lambda ratio.
* Must have received at least 2 or more lines of therapy, including a proteasome inhibitor (PI), an immunomodulatory imide (IMiD), and an anti-CD38 monoclonal antibody (mAb).
* Must be eligible to receive the Investigator's choice standard available therapy (SAT) based on approved prescribing information, previous MM treatment history, and institutional guidelines.

Exclusion Criteria:

* Clinically significant (per Investigator's judgment) drug or alcohol abuse within the last 6 months.
* Clinically significant conditions such as but not limited to the following: neurologic, psychiatric, endocrine, metabolic, immunologic, cardiovascular, pulmonary, or hepatic disease within the last 6 months that would adversely affect the participant's participation in the study.
* Central nervous system involvement of MM.
* Has received B-cell maturation antigen (BCMA)-targeted therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-05-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to Approximately 5 Years
  PFS is defined as the duration from the date of randomization to the date of confirmed disease progression (PD) determined by independent review committee (IRC) per international myeloma working group (IMWG) (2016) response criteria, or death, whichever occurs first.
Objective Response Rate (ORR) | Up to Approximately 5 Years
  ORR is defined as the percentage of participants who achieve confirmed partial response (PR) + VGPR + complete response (CR) + stringent complete response (sCR) or per IRC assessment.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to Approximately 5 Years
  OS is defined as the duration from the date of randomization to the date of the participant's death.
Change in Rate of Very Good Partial Response (VGPR) or Better (>= VGPR) | Up to Approximately 5 Years
  The rate of >= VGPR is defined as the proportion of participants who achieve a VGPR or better determined by IMWG (2016) response criteria, per IRC assessment, prior to the initiation of new myeloma therapy.
Change in Rate of CR or Better (>=CR) | Up to Approximately 5 Years
  >=CR is defined as the percentage of participants who achieve confirmed CR + sCR or per IRC assessment.
Change in Rate of Minimum Residual Disease (MRD) negativity with >= CR | Up to Approximately 5 Years
  MRD negativity with >= CR, defined as achievement of CR or better by IMWG (2016) response criteria (per IRC assessment) and MRD negative status as assessed by next-generation sequencing (NGS) Adaptive Clonoseq at 10^-5 threshold.
Change from Baseline in Disease Symptoms as Measured by the Disease Symptoms Domain of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Multiple Myeloma Module (EORTC QLQ-MY20) | Up to 6 Months
  The disease symptoms domain of EORTC QLQ-MY20 is a 6-item questionnaire to assess the physical function of the participant, with a higher score indicating a higher level of symptoms.
Change from Baseline in Physical Functioning as Measured by the Physical Functioning Domain of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) | Up to 6 Months
  The physical functioning domain of EORTC QLQ-C30 is a 5-item questionnaire to assess the physical function of the participant, with a higher score indicating worse functioning.
Time to Response (TTR) | Up to Approximately 5 Years
  TTR is defined as the number of months from the date of first dose to the date of best overall response of CR or PR ('responders') determined by IMWG criteria as assessed by IRC.
Duration of Response (DOR) | Up to Approximately 5 Years
  DOR is defined as the number of days from the day the response criteria are met to the date that disease progression as determined by the IRC.
Time-to-Progression (TTP) | Up to Approximately 5 Years
  TTP is defined as the number of days from the date of first dose to the date of earliest disease progression as determined by the IRC.
Time to Next Anti-lymphoma Therapy (TTNT) | Up to Approximately 5 Years
  TTNT is defined as the time from randomization to first documented administration of subsequent anti-lymphoma therapy.
Number of Participants with Event-free Survival (EFS) | Up to Approximately 5 Years
  EFS is defined as the time from randomization until adverse event determined by the IRC, or death, whichever occurs first.
Change from Baseline in Patient-Reported Outcomes Measurement Information System Fatigue Short Form 7a (PROMIS Fatigue SF 7a) | Up to Approximately 6 Months
  The PROMIS Fatigue SF7a is a 7-item short form that assesses the impact and experience of fatigue in the past 7 days. For each item, 5-point rating scales are used to measure frequency ("Never," "Rarely," "Sometimes," "Often," or "Always") with a higher score indicating a greater impact.
Change from Baseline in Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to Approximately 6 Months
  The PRO-CTCAE is a patient-reported outcome measurement system developed to assess symptomatic toxicity in participants in cancer clinical trials. PRO-CTCAE items are scored from 0 to 4 to evaluate common symptoms from study treatment on their frequency, severity, interference, amount, presence/absence.
Change from Baseline in Remaining Items in the EORTC QLQ-C30 | Up to Approximately 6 Months
  The EORTC QLQ-C30 assesses health-related quality of life in cancer patients participating in clinical trials. The EORTC QLQ-C30 comprises 5 functional scales (physical, role, emotional, social, cognitive), 8 single-item symptom scales (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, and dyspnea), as well as subscales assessing global health/quality of life and financial impact. Raw scores are transformed to a scale of 0 to 100, with higher scores representing better functioning/quality of life and greater symptom burden.
Change from Baseline in Remaining Items in the EORTC QLQ-MY20 | Up to Approximately 6 Months
  The EORTC QLQ-MY20 consists of four scales: two symptom scales (Disease Symptoms [6 items] and Side Effects of Treatment [10 items]), one function scale (Future Perspective [3 items]), and one single item (Body Image). Each item has four response options: "Not at all," "A little," "Quite a bit," or "Very much". All scores are then linearly transformed to a 0 to 100 scale. A higher score on the symptom scales indicates a higher level of symptoms, whereas higher scores on future perspective and body image indicate good functioning or support.
Change from Baseline in European Quality-of-Life 5-dimensional-5-level (EQ-5D-5L) | Up to Approximately 6 Months
  The EQ-5D-5L is a standardized, non-disease specific instrument used to measure health-related quality of life. The EQ-5D-5L assesses general health on 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/ depression). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems). The scores for the 5 dimensions are used to compute a single utility index score ranging from 0 to 1 representing the general health status of the individual, with higher scores indicating better health state.
Change from Baseline in Patient Global Impression of Severity (PGIS) | Up to Approximately 6 Months
  The self-report measure PGIS reflects a participant's belief about their lymphoma symptoms over the past 7 days. The PGIS is a 5-point scale depicting a participant's rating of overall severity.
Change from Baseline in Patient Global Impression of Change (PGIC) | Up to Approximately 6 Months
  The self-report measure PGIC reflects a participant's belief about the efficacy of treatment. The PGIC is a 7-point scale depicting a participant's rating of overall improvement since start of treatment. Participants rate their change as very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse.
Number of Participants with Skeletal-Related Event (SRE) | Up to Approximately 5 Years
  SREs are defined as the presence of any of the following spinal cord compression, pathologic fracture, surgery to bone, or radiation to bone.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (166):
- United States (46):
  - University of Alabama at Birmingham - Main /ID# 261434, Birmingham, Alabama
  - Mayo Clinic Hospital - Phoenix /ID# 263326, Phoenix, Arizona
  - Alta Bates Summit Medical Center for Research /ID# 261438, Berkeley, California
  - Providence - St. Jude Medical Center /ID# 262031, Fullerton, California
  - VA Loma Linda Healthcare System /ID# 261015, Loma Linda, California
  - Cedars-Sinai Medical Center /ID# 261008, Los Angeles, California
  - Rocky Mountain Cancer Centers - Lone Tree /ID# 278320, Lone Tree, Colorado
  - Mayo Clinic Hospital Jacksonville /ID# 263324, Jacksonville, Florida
  - Cancer Specialists of North Florida - Jacksonville - AC Skinner Parkway /ID# 246230, Jacksonville, Florida
  - Winship Cancer Institute of Emory University /ID# 262525, Atlanta, Georgia
  - University of Illinois Hospital and Health Sciences System /ID# 246349, Chicago, Illinois
  - Rush University Medical Center /ID# 265690, Chicago, Illinois
  - Nancy W. Knowles Cancer Center /ID# 271361, Elmhurst, Illinois
  - Springfield Clinic - First /ID# 262266, Springfield, Illinois
  - Our Lady Of The Lake Regional Medical Center /ID# 272780, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders-American Oncology Partners of Maryland /ID# 263637, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center /ID# 271535, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 261554, Boston, Massachusetts
  - Regents of the University of Michigan /ID# 261577, Ann Arbor, Michigan
  - Karmanos Cancer Institute - Detroit /ID# 266298, Detroit, Michigan
  - Henry Ford Hospital /ID# 262704, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute - McLaren Greater Lansing /ID# 259891, Lansing, Michigan
  - Mayo Clinic - Rochester /ID# 246228, Rochester, Minnesota
  - University of Missouri Hospital /ID# 261553, Columbia, Missouri
  - Nebraska Cancer Specialists - Omaha - Wright Street /ID# 276772, Omaha, Nebraska
  - New York Cancer & Blood Specialists - Bay Shore /ID# 261524, Bay Shore, New York
  - New York Cancer & Blood Specialists - Lake Success Medical Oncology /ID# 262953, New Hyde Park, New York
  - New York Cancer and Blood Specialists - New York /ID# 262951, New York, New York
  - Eastchester Center for Cancer Care /ID# 262952, The Bronx, New York
  - University of North Carolina /ID# 259854, Chapel Hill, North Carolina
  - Atrium Health Levine Cancer Institute /ID# 246199, Charlotte, North Carolina
  - Duke University Medical Center /ID# 259694, Durham, North Carolina
  - University Of Cincinnati Medical Center /ID# 246415, Cincinnati, Ohio
  - Cleveland Clinic Main Campus /ID# 246183, Cleveland, Ohio
  - Oregon Medical Research Center /ID# 262335, Portland, Oregon
  - Medical University of South Carolina /ID# 259692, Charleston, South Carolina
  - University of Tennessee Health Science Center /ID# 261622, Memphis, Tennessee
  - Baptist Memorial Hospital /ID# 270910, Memphis, Tennessee
  - The West Clinic /ID# 262444, Memphis, Tennessee
  - Vanderbilt University Medical Center /ID# 261621, Nashville, Tennessee
  - Oncology Consultants /ID# 276774, Houston, Texas
  - Texas Oncology - Northeast Texas /ID# 278304, Tyler, Texas
  - Virginia Cancer Specialists - Fairfax /ID# 262792, Fairfax, Virginia
  - Virginia Oncology Associates - Norfolk (Lake Wright) /ID# 278314, Norfolk, Virginia
  - VCU Massey Cancer Center: Dalton Oncology Clinic /ID# 261944, Richmond, Virginia
  - Northwest Medical Specialties Tacoma /ID# 276281, Tacoma, Washington
- Australia (7):
  - St George Hospital /ID# 261806, Kogarah, New South Wales
  - Liverpool Hospital /ID# 262159, Liverpool, New South Wales
  - Calvary Mater Newcastle /ID# 261804, Waratah, New South Wales
  - Princess Alexandra Hospital /ID# 261810, Woolloongabba, Queensland
  - Monash Health - Monash Medical Centre /ID# 262158, Clayton, Victoria
  - St Vincent's Hospital Melbourne /ID# 261808, Fitzroy Melbourne, Victoria
  - Box Hill Hospital /ID# 262784, Melbourne, Victoria
- Austria (4):
  - Universitaetsklinikum Krems /ID# 261509, Krems, Lower Austria
  - Medizinische Universitaet Graz /ID# 261908, Graz, Styria
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 245609, Linz, Upper Austria
  - Klinik Ottakring /ID# 245829, Vienna, Vienna
- Belgium (2):
  - Algemeen Ziekenhuis klina /ID# 260856, Brasschaat, Antwerpen
  - AZ Sint-Jan Brugge /ID# 245345, Bruges, West-Vlaanderen
- University Health Network_Princess Margaret Cancer Centre /ID# 261566, Toronto, Ontario, Canada
- China (18):
  - Beijing Chaoyang Hospital,Capital Medical University /ID# 245533, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital (East) - Dongdan Campus /ID# 245545, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital /ID# 245558, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center /ID# 245542, Guangzhou, Guangdong
  - People's Hospital of Henan Province /ID# 260918, Zhengzhou, Henan
  - Henan Cancer Hospital /ID# 245536, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 245549, Wuhan, Hubei
  - Zhongda Hospital Southeast University /ID# 245563, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University /ID# 245544, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 245537, Nanchang, Jiangxi
  - First Affiliated Hospital of China Medical University /ID# 245547, Shenyang, Liaoning
  - Second Affiliated Hospital of Xian Jiaotong University /ID# 261255, Xi'an, Shaanxi
  - Shanghai Tongji Hospital /ID# 245539, Shanghai, Shanghai Municipality
  - Institute of Hematology and Blood Diseases Hospital /ID# 265702, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital /ID# 260851, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 260883, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine /ID# 260882, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University /ID# 245550, Wenzhou, Zhejiang
- Czechia (4):
  - Fakultní Nemocnice Brno - Jihlavská /ID# 245689, Brno, Brno-mesto
  - Fakultní nemocnice Hradec Králové - Sokolská /ID# 245690, Hradec Králové, Hradec Kralove
  - Fakultni Nemocnice Ostrava /ID# 245686, Ostrava, Ostrava-mesto
  - Vseobecna Fakultni Nemocnice v Praze /ID# 245691, Prague, Praha 17
- Denmark (2):
  - Odense University Hospital /ID# 260924, Odense, Region Syddanmark
  - Vejle Sygehus /ID# 260923, Vejle, Region Syddanmark
- France (4):
  - Ch Saint Quentin /Id# 261856, Saint-Quentin, Aisne
  - Centre Hospitalier du Mans /ID# 261852, Le Mans, Sarthe
  - CH Henri Duffaut /ID# 261844, Avignon, Vaucluse
  - Centre Hospitalier Régional d'Orléans - Hôpital de la Source /ID# 261854, Orléans
- Germany (6):
  - Universitaetsklinikum Freiburg /ID# 262147, Freiburg im Breisgau, Baden-Wurttemberg
  - Staedtisches Klinikum Karlsruhe /ID# 272377, Karlsruhe, Baden-Wurttemberg
  - Klinikum Chemnitz - Flemmingstraße /ID# 273108, Chemnitz, Saxony
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 260689, Berlin
  - Centrum fuer Haematologie und Onkologie Bethanien /ID# 271982, Frankfurt am Main
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 260651, Hamburg
- Greece (4):
  - Alexandra General Hospital /ID# 240591, Athens, Attica
  - University General Hospital Attikon /ID# 240592, Athens, Attica
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 240596, Athens
  - General University Hospital of Thessaloniki AXEPA /ID# 240595, Thessaloniki
- Hungary (3):
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz /ID# 261648, Győr, Győr-Moson-Sopron
  - Semmelweis Egyetem /ID# 261647, Budapest
  - Del-pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet /ID# 261646, Budapest
- Israel (4):
  - Shaare Zedek Medical Center /ID# 245681, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 245497, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 245495, Tel Aviv, Tel Aviv
  - Rabin Medical Center. /ID# 245498, Petah Tikva
- Italy (5):
  - ASST Ovest Milanese /ID# 256813, Legnano, Milano
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 256808, Turin, Piedmont
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 256810, Rome, Roma
  - Azienda Ospedaliero Universitaria delle Marche /ID# 256812, Ancona
  - AOU Policlinico G. Rodolico - San Marco /ID# 256814, Catania
- Japan (17):
  - Anjo Kosei Hospital /ID# 263434, Anjo, Aichi-ken
  - Nagoya City University Hospital /ID# 263320, Nagoya, Aichi-ken
  - Chiba University Hospital /ID# 262006, Chiba, Chiba
  - University of Fukui Hospital /ID# 264222, Yoshida-gun, Fukui
  - Kyushu University Hospital /ID# 264704, Fukuoka, Fukuoka
  - Gifu Municipal Hospital /ID# 263321, Gifu, Gifu
  - Gunma University Hospital /ID# 262580, Maebashi, Gunma
  - Chugoku Central Hospital /ID# 263431, Fukuyama, Hiroshima
  - Hyogo Prefectural Amagasaki General Medical Center /ID# 265696, Amagasaki, Hyōgo
  - University Hospital Kyoto Prefectural University of Medicine /ID# 262585, Kyoto, Kyoto
  - Miyagi Cancer Center /ID# 265094, Natori-shi, Miyagi
  - Naha City Hospital /ID# 263972, Naha, Okinawa
  - The University of Osaka Hospital /ID# 263974, Suita-shi, Osaka
  - Saitama Prefectural Cancer Center /ID# 262586, Kitaadachi-gun, Saitama
  - Tokyo Metropolitan Komagome Hospital /ID# 277567, Bunkyo Ku, Tokyo
  - Japanese Red Cross Medical Center /ID# 261717, Shibuya-ku, Tokyo
  - University of Yamanashi Hospital /ID# 262912, Chuo-shi, Yamanashi
- Poland (3):
  - Uniwersytecki Szpital Kliniczny We Wroclawiu /ID# 260172, Wroclaw, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny Nr 1 w Lublinie /ID# 260168, Lublin, Lublin Voivodeship
  - Uniwersyteckie Centrum Kliniczne /ID# 260169, Gdansk, Pomeranian Voivodeship
- Portugal (3):
  - Fundacao Champalimaud /ID# 246258, Lisbon, Lisbon District
  - Unidade Local de Saude de Santa Maria, EPE /ID# 246255, Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE /ID# 246257, Porto
- Puerto Rico (2):
  - Hematology And Oncology Institute /ID# 272531, Manatí
  - Auxilio Mutuo Cancer Center /ID# 272565, San Juan
- South Africa (3):
  - Alberts Cellular Therapy /ID# 245725, Pretoria, Gauteng
  - Constantiaberg Haematology /ID# 261320, Cape Town, Western Cape
  - Haemalife Inc. /ID# 245724, Kuils River, Western Cape
- South Korea (5):
  - Seoul National University Hospital /ID# 245491, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 245492, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 245493, Seoul, Seoul Teugbyeolsi
  - Ulsan University Hospital /ID# 245490, Ulsan, Ulsan Gwang Yeogsi
  - Yonsei University Health System Severance Hospital /ID# 245489, Seoul
- Spain (6):
  - Instituto Catalan de Oncologia (ICO) Badalona /ID# 246398, Badalona, Barcelona
  - Complejo Hospitalario Universitario Ourense /ID# 246400, Ourense, Ourense
  - Hospital de Leon /ID# 261624, León
  - Hospital General Universitario Gregorio Maranon /ID# 246401, Madrid
  - Hospital Universitario de Salamanca /ID# 262218, Salamanca
  - Hospital Universitario y Politecnico La Fe /ID# 261625, Valencia
- Sweden (3):
  - Helsingborgs Lasarett /ID# 262513, Helsingborg, Skåne County
  - Uddevalla sjukhus /ID# 262034, Uddevalla, Västra Götaland County
  - Falu Lasarett /ID# 262231, Falun
- Taiwan (3):
  - National Taiwan University Hospital /ID# 245482, Taipei City, Taipei
  - China Medical University Hospital /ID# 245483, Taichung
  - Taichung Veterans General Hospital /ID# 261142, Taichung
- Turkey (Türkiye) (4):
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi /ID# 261672, Ankara
  - Antalya Egitim Ve Arastirma Hastanesi /ID# 261674, Antalya
  - Trakya University Medical Facu /ID# 261673, Edirne, Istanbul
  - Istanbul Florence Nightingale Hospital /ID# 271543, Şişli
- United Kingdom (7):
  - Addenbrookes Hospital /ID# 261104, Cambridge, Cambridgeshire
  - Western General Hospital - NHS Lothian /ID# 261106, Edinburgh, Edinburgh, City of
  - Dup_Guys and St Thomas NHS Foundation Trust - Guy's Hospital /ID# 262488, London, Greater London
  - Nottingham City Hospital /ID# 261105, Nottingham, Nottinghamshire
  - Leeds Teaching Hospitals NHS Trust /ID# 261101, Leeds, West Yorkshire
  - The Royal Marsden NHS Foundation Trust /ID# 262470, London
  - The Christie Hospital /ID# 261102, Manchester

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-574